CLINICAL TRIAL: NCT05469230
Title: Assessment of Cognitive Function, Fatigue and Health Related Quality of Life in Children With Beta Thalassemia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Elmorsi Abdelaziz Elderini Ibrahim, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/003783
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Change; Beta-Thalassemia; Fatigue; Quality of Life
MeSH Terms: conditions — beta-Thalassemia; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically developed children group: Typically developed children will be from both genders. the age range will be (8-16) years old and will be recruited from public governmental schools
- Beta thalassemia group: children diagnosed with beta thalassemia major and intermedia will be recruited from Abo-El-Rish Pediatric Hospital. the age will be (8-16) years and will be from both genders

SUMMARY:
This study aims to:

* Assess the cognitive function in children with beta thalassemia
* Evaluate the fatigue in beta thalassemic children
* Assess the health related quality of life measures in children with beta thalassemia.

DETAILED DESCRIPTION:
The cognitive abilities are extremely important for academic achievement. Despite their importance, the evaluation of cognitive function is rarely performed for thalassemia patients. So it is important to assess it and should be a routine comprehensive care of beta thalassemia patients to detect cases that suffer from verbal and performance dysfunction and subject them to the learning skills programs, so investigators can monitor any defects or problems that could arise early.

Thalassemia not only affect cognitive abilities, it has also many negative effects on physical health; the patients cannot perform activities easily, get fatigued easily and quickly. Also, emotional and social health aspects are affected. So, assessing health related quality of life is recognized as an indispensable indicator for a general evaluation of patients with thalassemia through which valuable evidence could be provided to improve treatments and to make effective decisions.

Cognitive function, fatigue and health related quality of life in children with beta thalassemia will be assessed by using valid and reliable scales. All the patients and controls will be subjected to assessment using the Arabic version of the Wechsler Intelligence Scale for Children which assess cognitive function and provide the output of the Verbal comprehension index ,Perceptual reasoning index, processing speed index, working memory index and a combined Full-Scale IQ test. The assessment included 15 subtests.

Health related quality of life will be assessed using the Arabic version of child proxy report of the Pediatric Quality of Life Inventory Generic Core Scale (version 4)( PedsQL). The PedsQL Inventory Generic Core Scales is a brief 23 items multidimensional instrument assessing the physical, emotional, social and school functioning domains. It is a reliable and valid tool designed to measure Health related quality of life The fatigue will be assessed using the Arabic version of child report of the Pediatric Quality of Life Inventory Multidimensional Fatigue Scale which covers three domains, including General Fatigue (6 items), Sleep/Rest Fatigue (6 items) and Cognitive Fatigue (6 items) .

Every child will be evaluated alone in spacious and quiet room free from any visual and auditory distractions.

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia group (Study group): Both genders will be included and their age range from 8 to 16 years old
* Typically developed children (control group):

  * Healthy children will be recruited from public governmental schools
  * Healthy controls, matching the patients in age, gender and educational level.
  * It will be ensured from their past medical history and clinical examination that they and their first-degree relatives never had any chronic disease, including thalassemia.
  * Both genders will be included
  * Their age range from 8 to 16 years old

Exclusion Criteria:

* Beta thalassemia group (study group): Any child Suffering from any other chronic diseases other than thalassemia

  • Having visual or auditory problems
* Typically developed children (control group):

any child suffering from medical illness, musculoskeletal deformities, visual and auditory problems.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Children diagnosed with beta thalassemia will be recruited from Abo El-Rish Pediatric Hospital .(Cairo University Hospitals)
  * Both genders will be included
  * Their age range from 8 to 16 years old shouldn't have any associated diseases with beta thalassemia
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
assessing the change in cognitive function | baseline to 6 months
  assessing the change in verbal comprehension, perceptual reasoning, processing speed, working memory and total IQ using Wecshler Intelligence Scale for Children (4th edition)
Assessing the change in fatigue | Baseline to 6 months
  assessing the change in General Fatigue,Sleep/Rest Fatigue and Cognitive Fatigue using Pediatric quality of life inventory multidimensional fatigue scale (child report)
Assessing the change in health related quality of life | Baseline to 6 months
  assessing the change in physical, emotional, social and school functioning domains using the Pediatric quality of life inventory Generic core scale (child report) (version 4)

CONTACTS AND LOCATIONS:
Overall Officials: Esraa ibrahim, M.Sc, Principal Investigator — Cairo University
Locations (1):
- Abo El-Rish Pediatric Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided